CLINICAL TRIAL: NCT06682312
Title: Element Boulder Clinical Investigation Plan Philips Non-Invasive Blood Pressure Validation Study
Brief Title: Philips Non-Invasive Blood Pressure Validation Study
Status: Terminated | Type: Observational
Why Stopped: Protocol violations resulting in wrong stratification requirements
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Element Materials Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: PR 2024-601
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Non Invasive Blood Pressure
Keywords: NIBP; Blood pressure; Spotcheck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pediatrics: Participants aged 3-12 years
  Interventions: Device: Non-invasive blood pressure
- Adults: Participants aged 12-85 years

INTERVENTIONS:
Device: Non-invasive blood pressure — Manual blood pressure via sphygmomanometer
  Or
  Non invasive blood pressure via earlyvue VS30 Monitor
  Groups: Pediatrics

SUMMARY:
The purpose of this study is to provide supporting documentation of the blood pressure performance for the Philips EarlyVue VS30 monitor on the intended adult and pediatric population. The same arm sequential method with dual observer auscultation will be used to collect data.

DETAILED DESCRIPTION:
The Philips EarlyVue VS30 monitor, and approved Philips Gentle Care cuffs will be evaluated in comparison to dual reference auscultation. The study will consist of a minimum of 85 participants, specifically, 35 children aged 3-12 years and 50 participants older than 12 years. The participants enrolled will approximate the distribution of blood pressures and biceps circumferences as outlined in ISO 81060-2:2018/AMD 2:2024. The maximum number of participants enrolled will not exceed 170 participants.

Blood pressure measurements will follow ISO 81060-2:2018/AMD 2:2024, Section 5.2.4.1 Same arm sequential method.

Two trained observers, typically a Registered Nurse (RN), Licensed Practical Nurse (LPN), or Respiratory Therapist (RT) will observe (listen to) the Korotkoff sounds at the artery at the site of cuff placement. The reference blood pressure measurements observed by the auscultators will be performed sequentially with the device under test. The auscultators will complete 1 or 2 initial baseline auscultatory reference blood pressure measurements and device under test measurements. This is followed by 3 to 8 paired blood pressure readings of auscultatory reference blood pressure measurements alternated with device under test measurements. All participants must contribute 3 valid paired data points requiring three DUT readings paired with three reference blood pressure readings. The reference blood pressure readings for analysis will be the average of the reference dual auscultation values before and after DUT reading.

The data included for the final analysis will contain no fewer than 35 participants aged 3-12 years, and no fewer than 50 participants over the age of 12 and a minimum of 255 valid paired observations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to provide an informed consent or have legally authorized representative consent to participate.
* Participants that are between 7 and 17 years of age must provide assent to participate in the study.
* Participant must be willing and able to comply with the study procedures.
* Participant or legally authorized representative must be able to read or write in English.
* Participant must be 3 to 85 years of age.
* Participants must have an arm circumference in the range of 14-45 centimeters.

Exclusion Criteria:

* Participant is unwilling to provide informed consent.
* Participants with deformities or abnormalities that may prevent proper application of the device under test.
* Participants whose upper arm circumference is less than 14 cm or greater than 45 cm.
* Female participants who are self-reported as pregnant, or who are self-reported as trying to get pregnant.
* Participants with known heart arrhythmias.
* Participants with peripheral vascular disease.
* Participants with clotting disorders.
* History of bleeding disorders or personal history of prolonged bleeding from injury
* History of blood clots
* Hemophilia
* Participants that cannot tolerate sitting for up to 1 hour.
* Participant with a blood pressure demographic that has already been filled.
* Other known health conditions that will prevent safe participation in the study upon disclosure in health assessment form or verbally.
* Participant is evaluated by the investigator or clinician and found to be medically unsuitable for participation in this study.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males and Females
Study Population: Healthy volunteers, both male and females aged 3-85. Minimum of 35 participants aged 3-12 and a minimum of 50 participants aged >12-85
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Validation of earlyvue VS30 Monitor | 2 weeks
  The primary objective of this study is to provide a validation following ISO 81060-2:2018/AMD 2:2024 for noninvasive blood pressure measurement accuracy for the Philips EarlyVue VS30 on the intended population. The EarlyVue VS30 will be compared to the reference sphygmomanometer via same arm sequential method with dual auscultators.
  The end goal is to pass the Criterion 1 and Criterion 2 of ISO 81060-2:2018/AMD 2:2024 Criterion 1
  * Mean Error of individual paired determinations ≤ ±5.0 mmHg
  * Standard Deviation of determination ≤ 8.0mmHg
  Criterion 2
  • Standard Deviation of the average paired determinations must meet the maximum permissible standard deviation in Table 1 - Averaged subject data acceptance (criterion 2) in mmHg per the standard

CONTACTS AND LOCATIONS:
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Study has been terminated and no analysis will be done